CLINICAL TRIAL: NCT06302569
Title: Activity of Pembrolizumab Plus Enfortumab Vedotin in Collecting Duct and Renal Medullary Carcinoma
Brief Title: Pembrolizumab Plus Enfortumab Vedotin in Collecting Duct and Renal Medullary Carcinoma
Acronym: REPRINT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giuseppe Procopio (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Procopio, Director of GenitoUrinary Oncology, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bellini INT 2024-511587-93-00
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Bellini Carcinoma; Collecting Duct Carcinoma; Renal Medullary Carcinoma
Keywords: Pembrolizumab; Enfortumab Vedotin; Non-clear cell renal cell carcinoma; Collecting Duct Carcinoma; Renal Medullary Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; enfortumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Enfortumab Vedotin (Experimental): Patients will be treated with Pembrolizumab q21 plus Enfortumab Vedotin 1,8q21 for 3 cycles (3 infusion of Pembrolizumab and 6 infusion of Enfortumab Vedotin) then radiological imaging will be repeated and patients with SD, PR or CR will continue pembrolizumab until disease progression, or unacceptable toxicities or completion of treatment (17 cycles). Patients with progressive disease after 3 cycles of study intervention will be treated as per clinical practice.
  Patients who will experience progressive disease during pembrolizumab monotherapy treatment could restart Enfortumab Vedotin.
  Interventions: Drug: Pembrolizumab + Enfortumab Vedotin

INTERVENTIONS:
Drug: Pembrolizumab + Enfortumab Vedotin — * Pembrolizumab will be given for a maximum of 2 years i.e. a total of 35 cycles of pembrolizumab with the q3 week dosing. Participants who complete study intervention after 2 years of pembrolizumab are eligible for up to 1 year of additional pembrolizumab (second course) upon experiencing disease progression.
  * Enfortumab Vedotin will be given for a maximum of 3 cycles on day 1 and day 3 each 3 weeks. EV treatment could be re-started in case of Progressive Disease RECIST v1.1 during pembrolizumab monotherapy treatment.
  Other Names: KEYTRUDA + PADCEV

SUMMARY:
This is a single-arm, monocentric, phase II trial, enrolling patients with histological diagnosis of collecting duct carcinoma and renal medullary carcinoma with locally advanced or metastatic disease who will be treated with Pembrolizumab plus Enfortumab Vedotin.

Approximately, 23 patients will be enrolled. At screening, pre-existing archival primary and metastatic FFPE tumor specimen will be collected and submitted for central pathology review and translational analysis. All participants will undergo baseline screening imaging for clinical staging. Patients will be treated with Pembrolizumab q21 plus Enfortumab Vedotin 1,8q21 for 3 cycles (3 infusion of Pembrolizumab and 6 infusion of Enfortumab Vedotin) then radiological imaging will be repeated and patients with SD, PR or CR will continue pembrolizumab until disease progression, unacceptable toxicities or completion of treatment (17 cycles). Patients with progressive disease after 3 cycles of study intervention will be treated as per clinical practice.

Patients who will experience progressive disease during pembrolizumab monotherapy treatment could restart Enfortumab Vedotin.

The study will also involve collection of a blood sample taken at the commencement of treatment, at the first cycle, after cycle 3 and at the end of treatment or progression of disease, to be used for research purposes.

DETAILED DESCRIPTION:
BACKGROUND Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD 1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2). Based on preclinical in vitro data, pembrolizumab has high affinity and potent receptor blocking activity for PD 1. Pembrolizumab has an acceptable preclinical safety profile and is in clinical development as an intravenous (IV) immunotherapy for advanced malignancies. Keytruda® (pembrolizumab) is indicated for the treatment of patients across a number of indications because of its mechanism of action to bind the PD-1 receptor on the T cell. For more details on specific indications refer to the Investigator brochure (IB).

Enfortumab Vedotin (EV) is an ADC comprised of a fully human anti-Nectin-4 IgG1 kappa mAb conjugated to the small molecule microtubule disrupting agent, MMAE, via a protease cleavable maleimidocaproyl vc linker. Conjugation takes place on cysteine residues that comprise the interchain disulfide bonds of the antibody to yield a product with a drug to antibody ratio of approximately 3:8.

EV binds to the V domain of Nectin-4 protein. In the presumed mechanism of action, the drug binds to the Nectin-4 protein on the cell surface and is internalized, causing proteolytic cleavage of the vc linker and intracellular release of MMAE. Free MMAE subsequently disrupts tubulin polymerization and leads to mitotic arrest.

PHARMACEUTICAL AND THERAPEUTIC BACKGROUND

Pembrolizumab. The importance of intact immune surveillance function in controlling outgrowth of neoplastic transformations has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T cells/FoxP3+ regulatory T-cells (T-regs) correlates with improved prognosis and long-term survival in solid malignancies, such as ovarian, colorectal, and pancreatic cancer; hepatocellular carcinoma; malignant melanoma; and renal cell carcinoma. Tumor-infiltrating lymphocytes can be expanded ex vivo and reinfused, inducing durable objective tumor responses in cancers such as melanoma.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an immunoglobulin (Ig) superfamily member related to cluster of differentiation 28 (CD28) and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) that has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD L1 and/or PD-L2).

The structure of murine PD-1 has been resolved. PD-1 and its family members are type I transmembrane glycoproteins containing an Ig-variable-type (IgV type) domain responsible for ligand binding and a cytoplasmic tail responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif, and an immunoreceptor tyrosine-based switch motif. Following T-cell stimulation, PD-1 recruits the tyrosine phosphatases, SHP-1 and SHP-2, to the immunoreceptor tyrosine-based switch motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3 zeta (CD3ζ), protein kinase C-theta (PKCθ), and zeta-chain-associated protein kinase (ZAP70), which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down-modulates T cell responses is similar to, but distinct from, that of CTLA-4, because both molecules regulate an overlapping set of signaling proteins. As a consequence, the PD 1/PD-L1 pathway is an attractive target for therapeutic intervention in Collecting Duct Carcinoma and Renal Medullary Carcinoma.

Enfortumab Vedotin Nectin-4 is a 66 kDa type I transmembrane protein that belongs to the Nectin family of adhesion molecules. It is composed of an ECD containing 3 Ig-like subdomains, a transmembrane helix, and an intracellular region. Nectins are thought to mediate Ca2+-independent cell-cell adhesion via both homophilic and heterophilic trans- interactions at adherens junctions where they can recruit cadherins and modulate cytoskeletal rearrangements. Sequence identity of Nectin-4 to other Nectin family members is low and ranges from 25% to 30% in the ECD.

The 3 Ig-like subdomains in the ECD of Nectin-4 are designated V, C1, and C2. The C1 domain is responsible for cisplatin-interaction (homodimerization), while V domains of most Nectin molecules contribute to trans-interaction and cell-cell adhesion.

Nectin-4 was originally identified by bioinformatics and cloned from human trachea. In humans, Nectin-4 is normally expressed in keratinocytes of the skin, sweat glands, hair follicles, transitional epithelium of the bladder, salivary gland ducts, esophagus, breast, and stomach. Nectin-4 was identified as markedly upregulated in urothelial carcinoma using suppression subtractive hybridization on a pool of urothelial carcinoma specimens. Immunohistochemical characterization of expression in multiple tumor specimens demonstrated high levels of Nectin-4 in bladder, breast, pancreatic, lung, ovarian and other cancers.

Enfortumab Vedotin in Combination with Pembrolizumab. Combining PD-1/PD-L1 inhibitors with a novel therapy, such as EV, may improve patient outcomes. Data from preclinical studies of brentuximab vedotin (a CD30-directed ADC comprising the same linker and MMAE payload as EV), shows potential to induce ICD, antigen presentation, and tumor immune infiltration. These results suggest that the effects are due to MMAE. Treatment with brentuximab vedotin in vitro and in preclinical models has been shown to induce hallmarks of ICD. ICD is characterized by induction of the endoplasmic reticulum stress response and subsequent surface presentation of DAMPs immune stimulatory molecules. These DAMPs induce innate immune migration and activation into the tumor microenvironment.

Based on the potential enhancement of immune response, it is hypothesized that combining EV with pembrolizumab will result in improved response leading to prolonged PFS and OS in patients with Collecting Duct Carcinoma and Renal Medullary Carcinoma with minimal overlapping toxicities between the 2 agents.

RATIONALE FOR THE TRIAL AND SELECTED POPULATION Non-clear cell renal cell carcinomas (nccRCC) comprise several rare and poorly described diseases. Among them, Renal medullary carcinoma (RMNC) represents less than 0,5% and Collecting Duct Carcinoma (CDC) represents 1% of all renal cell carcinomas. Both are characterized by an aggressive clinical behaviour and a particular poor prognosis. Both tumors are under-represented in prospective randomized trials predominantly including clear-cell histotype. Thus, a standard of treatment for these rare and aggressive histologies has not been defined yet. Based on the data of a small phase II study with responses of 23%, the more used first line therapy in both cases is a platinum-based cytotoxic chemotherapy that has the ability to control the disease but only for a limited time. More recently, the prospective BONSAI trial met its primary endpoint showing encouraging efficacy of cabozantinib in first line with an objective response (ORR) of 35% in 25 patients with metastatic CDC (mCDC). Immune-checkpoint inhibitors (ICI) such as Pembrolizumab in combination with Tyrosine Kinase Inhibitors are now recommended as standard-of-care options for clear-cell renal cell carcinoma due to the relevant results in term of antitumor activity and Overall Survival (OS). Cases of excellent response to ICI are reported in literature also in previously treated mCDC patients. Enfortumab Vedotin showed encouraging activity in different tumour types and when combined with pembrolizumab showed relevant results in term of ORR and PFS. More recently, the combination of EV and pembrolizumab in the EV-103/KEYNOTE-869 (NCT03288545) study has demonstrated dramatic improvement in ORR in cisplatin- ineligible patients with locally advanced and metastatic urothelial carcinoma, with a preliminary ORR of 73% (95% CI: 58, 85) regardless of PD-L1 expression level.

Due to the mechanism of action of Enfortumab Vedotin, the expression of NECTIN-4 in CDC is under analysis in the CICERONE trial (NCT05372302). Unpublished results from this trial, state that NECTIN-4 is expressed in 30% of CDC tissue. Furthermore, biology of CDC and of Urothelial Carcinoma is similar, and this support the expression of NECTIN-4 in this orphan disease and the activity of EV.

Based on the encouraging data regarding the use of ICI in clear cell renal cell carcinoma, the investigators hypothesize that in these histotypes it may be useful to evaluate in more depth the action of drugs that act on the immune system in combination with Antibody-Drug Conjugate (ADC).

PLANNED EXPLORATORY BIOMARKER RESEARCH Analysis on biomarkers is exploratory by nature and will be performed retrospectively after the main study analysis is completed. Tissue assessments will include the identification of somatic mutations in CDC and the assessment of the mutational load by focused exome analysis, as well as the identification of transcript fusions by RNA sequencing.

Plasma and viable peripheral blood mononuclear cell (PBMC) will be isolated and stored frozen for subsequent analysis. PBMC will be studied for immune cell profile by multicolor cytofluorimetry (including frequency and activation state of antitumor and immunosuppressive cell subsets of both innate and adaptive immunity), associated with gene-expression profiling and Cibersort analysis for assessing the activation state of the immune cell subsets.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic or advanced Collecting Duct Carcinoma or Medullary Renal Cell Carcinoma will be enrolled in this study.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have confirmed histology diagnosis of Collecting Duct Carcinoma or Medullary Renal Cell Carcinoma by central pathology review.
* Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 10 days prior to the start of study intervention.
* Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

Hepatitis B screening tests are not required unless:

1. Known history of HBV infection
2. As mandated by local health authority

   * Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.

Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Hepatitis C screening tests are not required unless:

a) Known history of HCV infection b) As mandated by local health authority

* HIV-infected participants must have well-controlled HIV on ART, defined as:

  1. Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening
  2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
  3. It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
  4. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study
  5. The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)

     Exclusion Criteria:
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy, including investigational agents, within 2 weeks prior to treatment allocation.
* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS diseases permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
ORR in patients treated with Pembrolizumab plus Enfortumab Vedotin | 24 Months
  The proportion of patients who have a partial or complete response to Pembrolizumab + Enfortumab Vedotin

SECONDARY OUTCOMES:
Progression-free survival (PFS) in patients treated with Pembrolizumab plus Enfortumab Vedotin | 24 Months
  The time from assignment to Pembrolizumab plus Enfortumab Vedotin to disease progression or death from any cause
Overall-survival (OS) in patients treated with Pembrolizumab plus Enfortumab Vedotin | 48 Months
  Survival from assignment to Pembrolizumab plus Enfortumab Vedotin to time of death.
Number of Participants treated with Pembrolizumab + Enfortumab Vedotin who experience AEs/SAEs | 24 Months
  The incidence of, causality, and outcome of AEs/SAEs. AEs will be assessed as defined by CTCAE, Version [5.0].

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy
Locations (1):
- Fondazione Irccs Istituto Dei Tumori Di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Procopio G, Sepe P, Claps M, Buti S, Colecchia M, Giannatempo P, Guadalupi V, Mariani L, Lalli L, Fuca G, de Braud F, Verzoni E. Cabozantinib as First-line Treatment in Patients With Metastatic Collecting Duct Renal Cell Carcinoma: Results of the BONSAI Trial for the Italian Network for Research in Urologic-Oncology (Meet-URO 2 Study). JAMA Oncol. 2022 Jun 1;8(6):910-913. doi: 10.1001/jamaoncol.2022.0238. PMID 35420628
- [Result] Oudard S, Banu E, Vieillefond A, Fournier L, Priou F, Medioni J, Banu A, Duclos B, Rolland F, Escudier B, Arakelyan N, Culine S; GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales). Prospective multicenter phase II study of gemcitabine plus platinum salt for metastatic collecting duct carcinoma: results of a GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales) study. J Urol. 2007 May;177(5):1698-702. doi: 10.1016/j.juro.2007.01.063. PMID 17437788
- [Result] Pagani F, Colecchia M, Sepe P, Apollonio G, Claps M, Verzoni E, de Braud F, Procopio G. Collecting ducts carcinoma: An orphan disease. Literature overview and future perspectives. Cancer Treat Rev. 2019 Sep;79:101891. doi: 10.1016/j.ctrv.2019.101891. Epub 2019 Aug 27. PMID 31491662
- [Result] Challita-Eid PM, Satpayev D, Yang P, An Z, Morrison K, Shostak Y, Raitano A, Nadell R, Liu W, Lortie DR, Capo L, Verlinsky A, Leavitt M, Malik F, Avina H, Guevara CI, Dinh N, Karki S, Anand BS, Pereira DS, Joseph IB, Donate F, Morrison K, Stover DR. Enfortumab Vedotin Antibody-Drug Conjugate Targeting Nectin-4 Is a Highly Potent Therapeutic Agent in Multiple Preclinical Cancer Models. Cancer Res. 2016 May 15;76(10):3003-13. doi: 10.1158/0008-5472.CAN-15-1313. Epub 2016 Mar 24. PMID 27013195
- [Result] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Result] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Result] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Result] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Result] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Result] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Result] Takai Y, Ikeda W, Ogita H, Rikitake Y. The immunoglobulin-like cell adhesion molecule nectin and its associated protein afadin. Annu Rev Cell Dev Biol. 2008;24:309-42. doi: 10.1146/annurev.cellbio.24.110707.175339. PMID 18593353
- [Result] Rikitake Y, Takai Y. Interactions of the cell adhesion molecule nectin with transmembrane and peripheral membrane proteins for pleiotropic functions. Cell Mol Life Sci. 2008 Jan;65(2):253-63. doi: 10.1007/s00018-007-7290-9. PMID 17928952
- [Result] Wahler D, Reymond JL. Novel methods for biocatalyst screening. Curr Opin Chem Biol. 2001 Apr;5(2):152-8. doi: 10.1016/s1367-5931(00)00184-8. PMID 11282341
- [Result] Takai Y, Miyoshi J, Ikeda W, Ogita H. Nectins and nectin-like molecules: roles in contact inhibition of cell movement and proliferation. Nat Rev Mol Cell Biol. 2008 Aug;9(8):603-15. doi: 10.1038/nrm2457. PMID 18648374
- [Result] Fabre-Lafay S, Monville F, Garrido-Urbani S, Berruyer-Pouyet C, Ginestier C, Reymond N, Finetti P, Sauvan R, Adelaide J, Geneix J, Lecocq E, Popovici C, Dubreuil P, Viens P, Goncalves A, Charafe-Jauffret E, Jacquemier J, Birnbaum D, Lopez M. Nectin-4 is a new histological and serological tumor associated marker for breast cancer. BMC Cancer. 2007 May 2;7:73. doi: 10.1186/1471-2407-7-73. PMID 17474988
- [Result] Rosenberg J, Sridhar SS, Zhang J, Smith D, Ruether D, Flaig TW, Baranda J, Lang J, Plimack ER, Sangha R, Heath EI, Merchan J, Quinn DI, Srinivas S, Milowsky M, Wu C, Gartner EM, Zuo P, Melhem-Bertrandt A, Petrylak DP. EV-101: A Phase I Study of Single-Agent Enfortumab Vedotin in Patients With Nectin-4-Positive Solid Tumors, Including Metastatic Urothelial Carcinoma. J Clin Oncol. 2020 Apr 1;38(10):1041-1049. doi: 10.1200/JCO.19.02044. Epub 2020 Feb 7. PMID 32031899
- [Result] Gargiuli C, Sepe P, Tessari A, Sheetz T, Colecchia M, de Braud FGM, Procopio G, Sensi M, Verzoni E, Dugo M. Integrative Transcriptomic Analysis Reveals Distinctive Molecular Traits and Novel Subtypes of Collecting Duct Carcinoma. Cancers (Basel). 2021 Jun 10;13(12):2903. doi: 10.3390/cancers13122903. PMID 34200770
- [Result] Buti S, Trentini F, Sepe P, Claps M, Isella L, Verzoni E, Procopio G. BONSAI-2 study: Nivolumab as therapeutic option after cabozantinib failure in metastatic collecting duct carcinoma patients. Tumori. 2023 Aug;109(4):418-423. doi: 10.1177/03008916221141483. Epub 2022 Dec 6. PMID 36474412
- [Result] Procopio G, Verzoni E, Iacovelli R, Colecchia M, Torelli T, Mariani L. Is there a role for targeted therapies in the collecting ducts of Bellini carcinoma? Efficacy data from a retrospective analysis of 7 cases. Clin Exp Nephrol. 2012 Jun;16(3):464-7. doi: 10.1007/s10157-012-0589-3. Epub 2012 Jan 26. PMID 22278601
- [Result] Mennitto A, Verzoni E, Peverelli G, Alessi A, Procopio G. Management of Metastatic Collecting Duct Carcinoma: An Encouraging Result in a Patient Treated With Cabozantinib. Clin Genitourin Cancer. 2018 Jun;16(3):e521-e523. doi: 10.1016/j.clgc.2018.03.010. Epub 2018 Mar 27. No abstract available. PMID 29656939